CLINICAL TRIAL: NCT06169124
Title: A Phase II Study of Androgen Receptor (AR) Inhibition by Darolutamide in Combination With Leuprolide Acetate and Exemestane in Recurrent Adult-Type Ovarian Granulosa Cell Tumor
Brief Title: Study to Test the Drug Darolutamide Along With the Drugs Leuprolide Acetate and Exemestane in Patients With Recurrent Ovarian Granulosa Cell Tumors
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2023-06524; NCI-2023-06524 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NRG-GY033 (Other: NRG Oncology); NRG-GY033 (Other: CTEP); U10CA180868 (NIH)
Record Dates: First submitted 2023-12-07; First posted 2023-12-13 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-12

CONDITIONS: Adult Ovarian Granulosa Cell Tumor
MeSH Terms: conditions — Granulosa cell tumor of the ovary | interventions — Specimen Handling; X-Rays; darolutamide; exemestane; Leuprolide; luprolide acetate gel depot; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (exemestane, darolutamide, leuprolide acetate) (Experimental): Patients receive exemestane PO QD and darolutamide PO BID starting on days -14 to -7 prior to C1D1 and then on days 1-28 of each cycle. Patients receive leuprolide acetate IM on day 1 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo chest CT or chest x-ray and CT, MRI, or PET/CT as well as blood sample collection throughout the study. Patients undergo collection of archived tissue during screening.
  Interventions: Procedure: Biospecimen Collection; Procedure: Chest Radiography; Procedure: Computed Tomography; Drug: Darolutamide; Drug: Exemestane; Drug: Leuprolide Acetate; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo archived tissue and blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Chest Radiography — Undergo chest x-ray
  Other Names: Chest X-ray
Procedure: Computed Tomography — Undergo CT and/or PET/CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Drug: Darolutamide — Given PO
  Other Names: Antiandrogen ODM-201; BAY 1841788; BAY-1841788; BAY1841788; Nubeqa; ODM 201; ODM-201; ODM201
Drug: Exemestane — Given PO
  Other Names: Aromasin; FCE-24304
Drug: Leuprolide Acetate — Given IM
  Other Names: A 43818; A-43818; A43818; Abbott 43818; Abbott-43818; Carcinil; Depo-Eligard; Eligard; Enanton; Enantone; Enantone-Gyn; Fensolvi; Ginecrin; LEUP; Leuplin; Leuprorelin Acetate; Lucrin; Lucrin Depot; Luprodex Depot; Lupron; Lupron Depot; Lupron Depot-3 Month; Lupron Depot-4 Month; Lupron Depot-Ped; Lutrate; Procren; Procrin; Prostap; TAP 144; TAP-144; TAP144; Trenantone; Uno-Enantone; Viadur
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT

SUMMARY:
This phase II trial tests how well darolutamide in combination with leuprolide acetate and exemestane works in treating patients with ovarian granulosa cell tumors that have come back after a period of improvement (recurrent). Darolutamide is in a class of medications called androgen receptor inhibitors. It works by blocking the effects of androgen (a male reproductive hormone) to stop the growth and spread of tumor cells. Leuprolide acetate is in a class of medications called gonadotropin-releasing hormone agonists. It works by decreasing the amount of certain hormones in the body. Exemestane is in a class of medications called aromatase inhibitors which has anti-estrogen and anticancer activities. Exemestane binds to and inhibits the enzyme aromatase, thereby blocking the conversion of androgens to estrogens. This lowers estrogen levels in the blood circulation causing the tumor cells to grow more slowly or stop growing completely. The combination of darolutamide, leuprolide acetate, and exemestane may be an effective approach to shrinking or stabilizing recurrent ovarian granulosa cell tumors or preventing them from coming back.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the objective response rate of darolutamide, leuprolide acetate, and exemestane in recurrent adult-type granulosa cell tumors of the ovary (AGCT).

SECONDARY OBJECTIVES:

I. To determine duration of response of darolutamide, leuprolide acetate, and exemestane in recurrent adult-type granulosa cell tumors of the ovary (AGCT).

II. To determine progression-free survival of darolutamide, leuprolide acetate, and exemestane when used in recurrent adult-type granulosa cell tumors of ovary (AGCT).

III. To determine overall survival of darolutamide, leuprolide acetate, and exemestane when used in recurrent adult-type granulosa cell tumors of ovary (AGCT).

IV. To elucidate the toxicities of darolutamide, leuprolide acetate, and exemestane when used in recurrent adult-type granulosa cell tumors of ovary (AGCT).

EXPLORATORY OBJECTIVE:

I. To determine biomarkers predictive of response to darolutamide, leuprolide acetate, and exemestane.

OUTLINE:

Patients receive exemestane orally (PO) once daily (QD) and darolutamide PO twice daily (BID) starting on days -14 to -7 prior to cycle 1, day 1 (C1D1) and then on days 1-28 of each cycle. Patients receive leuprolide acetate intramuscularly (IM) on day 1 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo chest computed tomography (CT) or chest x-ray and CT, magnetic resonance imaging (MRI), or positron emission tomography (PET)/CT as well as blood sample collection throughout the study. Patients undergo collection of archived tissue during screening.

Upon completion of study treatment, patients are followed up every 3 months for 2 years and then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Physicians should consider the following when evaluating if the patient is appropriate for this protocol:

  * Patients must have adequate health that permits completion of the study requirements and required follow up
  * For patients with known human immunodeficiency virus (HIV), hepatitis B virus (HBV), and/or hepatitis C virus (HCV) infection:

    * HIV-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial
    * For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
    * Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
  * Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial

In addition:

* The effects of the combination of darolutamide, leuprolide acetate, and exemestane on the developing human fetus are unknown. For this reason, and because androgen receptor inhibitor agents as well as other therapeutic agents used in this trial are known to be teratogenic, participants of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) during study therapy and for 1 month following the completion of study therapy. Should a participant become pregnant or suspect pregnancy while participating in this study, they should inform their treating physician immediately

  * Submission of tissue is required. Investigators should check with their pathology department regarding release of tissue before approaching patients about participation in the trial
  * Histologically confirmed diagnosis of recurrent adult-type granulosa cell tumor
  * Patient must have measurable disease. Measurable disease is defined in the protocol per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria. Measurable disease is defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded). Each lesion must be ≥ 10 mm when measured by CT or MRI. Lymph nodes must be ≥ 15 mm in short axis when measured by CT or MRI
  * Patient must have had ≥1 treatment regimen
  * Subject must have progressed on an aromatase inhibitor (letrozole, exemestane, anastrozole) in a prior treatment line
  * Age ≥ 18 years
  * Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2
  * Not pregnant and not nursing
  * Absolute neutrophil count (ANC) ≥ 1,500 cells/mm^3
  * Platelets ≥ 100,000 cells/mm^3
  * Hemoglobin ≥ 8 g/dl
  * Creatinine clearance (CrCL) of ≥ 30 mL/min by the Cockcroft-Gault formula
  * Total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN) (patients with known Gilbert's disease who have bilirubin level ≤ 3 x ULN may be enrolled)
  * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 1.5 x institutional ULN
  * Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class 2B or better
  * No active infection requiring parenteral antibiotics
  * Patients with current evidence of intra-abdominal abscess, abdominal/pelvic fistula (not diverted), gastrointestinal perforation, gastrointestinal (GI) obstruction, and/or need for drainage nasogastric or gastrostomy tube
  * The patient or a legally authorized representative must provide study-specific informed consent prior to study entry and, for patients treated in the United States (U.S.), authorization permitting release of personal health information

Exclusion Criteria:

* Prior treatment with AR inhibitors
* Known hypersensitivity to the study drugs or their ingredients

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2024-02-08 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | Within 9 months of initiating study treatment
  Defined as a complete response (CR) or partial response (PR) as assessed by Response Evaluation Criteria in Solid Tumors version 1.1 criteria. Exact 95% confidence limits, accounting for interim analysis, will be provided in the final report.

SECONDARY OUTCOMES:
Duration of response | From the time measurement criteria are met for CR or PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented, assessed up to 5 years
  Median duration of response with a corresponding 95% confidence interval will be estimated. The duration of overall CR is measured from the time measurement criteria are first met for CR until the first date that progressive disease is objectively documented. Stable disease is measured from the start of the treatment until the criteria for progression are met, taking as reference the smallest measurements recorded since date of study entry, including the baseline measurements.
Progression-free survival (PFS) | From study entry to time of progression or death, whichever occurs first, or date of last contact with known progression free status if neither progression nor death has occurred, assessed up to 5 years
  Will be graphed using Kaplan-Meier methods. Median PFS will be estimated with corresponding 95% confidence intervals.
Overall survival (OS) | From study entry to time of death or the date of last contact, assessed up to 5 years
  Will be graphed using Kaplan-Meier methods. Median OS will be estimated with corresponding 95% confidence intervals.
Incidence of adverse events | Up to 5 years
  Common Terminology Criteria for Adverse Events version 5 will be used to grade and categorize adverse events. Safety will be assessed beginning with the initial dose of any treatment. Descriptive statistics, including frequencies of maximum grade of adverse events by term and category will be reported. Adverse events categorized as grade 5 will be individually reported.

OTHER OUTCOMES:
Biomarkers predictive of response | Up to 5 years
  Local estrogen receptor and progesterone receptor immunohistochemistry results will be examined as possible predictive biomarkers of response to darolutamide, leuprolide acetate, and exemestane.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Hopp, Principal Investigator — NRG Oncology
Locations (66):
- United States (66):
  - Cedars Sinai Medical Center, Los Angeles, California
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Saint Alphonsus Cancer Care Center-Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Clinic Cancer Services - Sandpoint, Sandpoint, Idaho
  - Northwestern University, Chicago, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Northwestern Medicine Cancer Center Kishwaukee, DeKalb, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - Northwestern Medicine Grayslake Outpatient Center, Grayslake, Illinois
  - Northwestern Medicine Lake Forest Hospital, Lake Forest, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Northwestern Medicine Orland Park, Orland Park, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Ascension Saint Vincent Indianapolis Hospital, Indianapolis, Indiana
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - MaineHealth Maine Medical Center- Scarborough, Scarborough, Maine
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - University of Michigan Rogel Cancer Center, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Brighton, Brighton, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Canton, Canton, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Chelsea Hospital, Chelsea, Michigan
  - Cancer Hematology Centers - Flint, Flint, Michigan
  - Genesee Hematology Oncology PC, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Trinity Health Grand Rapids Hospital, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Beacon Kalamazoo Cancer Center, Kalamazoo, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Trinity Health Muskegon Hospital, Muskegon, Michigan
  - Cancer and Hematology Centers of Western Michigan - Norton Shores, Norton Shores, Michigan
  - Corewell Health Reed City Hospital, Reed City, Michigan
  - Corewell Health Lakeland Hospitals - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - University of Michigan Health - West, Wyoming, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology Ann Arbor Campus, Ypsilanti, Michigan
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Community Medical Center, Missoula, Montana
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Atrium Health Cabarrus/LCI-Concord, Concord, North Carolina
  - Miami Valley Hospital South, Centerville, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Saint Alphonsus Cancer Care Center-Ontario, Ontario, Oregon
  - Legacy Good Samaritan Hospital and Medical Center, Portland, Oregon
  - Legacy Meridian Park Hospital, Tualatin, Oregon
  - Legacy Salmon Creek Hospital, Vancouver, Washington
  - West Virginia University Charleston Division, Charleston, West Virginia
  - ThedaCare Regional Cancer Center, Appleton, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm